CLINICAL TRIAL: NCT00373165
Title: Open, Randomised Study Comparing Preemptive Therapy With Intravenous Ganciclovir With and Without Additional Oral Ganciclovir for CMV Prophylaxis in Immunosuppressed Renal Transplant Patients Receiving Monitoring of CMV Viral Load
Brief Title: Prophylaxis With Ganciclovir Improves Graft Survival in Renal Allograft Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lower Saxony Center for Nephrology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ML19827
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: DNA Virus Infection; Herpesviridae Infections; Cytomegalovirus Infection
Keywords: Renal Transplantation; CMV; Ganciclovir; Prophylaxis; Preemptive Therapy; Graft Survival; Proteomics
MeSH Terms: conditions — DNA Virus Infections; Herpesviridae Infections; Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
Study Phase: IV

Study Type: Open-label, multicenter, randomised clinical trial with two arms stratified for an intensified immunosuppressive regimen in patients at high risk for acute rejection.

Study Description: 148 kidney transplant recipients at risk for CMV disease were randomized and treated with ganciclovir capsules for 3 months (Group A, prophylaxis, N=74) or received ganciclovir IV only in case of proven CMV viral load (Group B, preemptive therapy, N=74). Initially, a 2 months follow up was planned in this trial. However, the study group decided to offer a longterm follow up to all patients and amended the protocol, respectively.

The aim of the study was to identify the most efficacious way to prevent renal transplant recipients from CMV disease and to find out, if one of these two strategies may increase graft or patient survival. Therefore, both wellknown approaches of CMV prevention were compared in two study groups:

Prophylaxis (Group A): Oral primary prophylaxis with ganciclovir capsules was started directly after transplantation and performed until day 90. In case of CMV infection (proven CMV viral load) or symptomatic CMV disease, treatment with ganciclovir IV was initiated.

Preemptive Therapy (Group B): No oral primary prophylaxis was given. Treatment with ganciclovir IV was given to patients with proven CMV viral load (CMV infection or CMV disease) only.

DETAILED DESCRIPTION:
Disease Background: More than 60 % of adult people are asymptomatically infected with cytomegalovirus (CMV). Due to immunosuppressive therapy, renal graft recipients are at risk for CMV infection and life-threatening disease. CMV can cause a variety of symptoms in the immunocompromised host, including CMV retinitis, pneumonia or colitis. After grafting, CMV disease most commonly occurs in the transplanted organ and can trigger graft dysfunction and acute rejection. Therefore, prophylaxis or preemptive therapy should be used in order to prevent graft recipients from CMV disease.

* CMV prophylaxis means the administration of antiviral agents to all patients at risk for CMV disease, directly after transplantation, i.e. for 3 months. Prophylaxis is in particular used for patients at high risk for CMV disease.
* CMV preemptive therapy (or targeted prophylaxis) means CMV monitoring and initiation of induction therapy with antiviral agents in patients with proven CMV viral load only (CMV infection). This prevents non-infected patients from being exposed to antiviral drugs and the related side effects like neutropenia or renal toxicity. Preemptive therapy is in particular used for patients at lower or moderate risk for CMV disease.

Study Description: 148 kidney transplant recipients at risk for CMV disease were randomized and treated with ganciclovir capsules for 3 months (Group A, prophylaxis, N=74) or received ganciclovir IV only in case of proven CMV viral load (Group B, preemptive therapy, N=74). Initially, a 2 months follow up was planned in this trial. However, the study group decided to offer a longterm follow up to all patients and amended the protocol, respectively.

The aim of the study was to identify the most efficacious way to prevent renal transplant recipients from CMV disease and to find out, if one of these two strategies may increase graft or patient survival. Therefore, both wellknown approaches of CMV prevention were compared in two study groups:

Prophylaxis (Group A): Oral primary prophylaxis with ganciclovir capsules was started directly after transplantation and performed until day 90. In case of CMV infection (proven CMV viral load) or symptomatic CMV disease, treatment with ganciclovir IV was initiated.

Preemptive Therapy (Group B): No oral primary prophylaxis was given. Treatment with ganciclovir IV was given to patients with proven CMV viral load (CMV infection or CMV disease) only.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients after living or postmortal donation
* CMV seropositive donor or recipient of the kidney transplant: D+/R-, D+/R+ or D-/R+
* Laboratory parameters: 50.000/ml thrombocytes and/or 1000/ml neutrophils
* Immunosuppression including MMF

Main Exclusion Criteria:

* Woman who are pregnant, breastfeeding or using unreliable birth control methods
* Forbidden concomitant medications during the 12 month observation period of the study are:
* Virustatic drugs, active against CMV: Foscarnet, Cidofovir (HPMPC), Acyclovir, Valaciclovir, Famciclovir/Penciclovir, Lobucavir, Antisense compound
* Antimetabolites: Fluorouracil, Mercaptopurine, Methotrexate, Thioguanine, Hydroxurea
* Alkylating substances: Busulfan, Carmustine, Chlorambucil, Cisplatin, Cyclophosphamide, Dacarbazine (DTIC), Lomustine, Mechlormethamine, Melphalan, Streptozotocin, Tiothepa, Uracil mustard
* anti CMV immunoglobulins (except in the case of signs of CMV infection) such as anti CMV hyperimmunoglobulins and immunoglobulins
* Known hypersensitivity to ganciclovir
* Patients with active CMV infection or positive viraemia at randomization
* Severe gastro-intestinal diseases which may interfere with the oral resorption of ganciclovir
* Conversion of immunosuppression (Replacement of MMF)
* Participation in another clinical drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-08; Study Completion 2003-10

PRIMARY OUTCOMES:
The impact of CMV infection on graft function, incidence of CMV infection and creatinine clearance in both study groups at month 12. long-term graft and patient survival. Neutrophil counts and creatinine clearance were measured on a regular basis.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Kliem, MD, Study Chair — Lower Saxony Center for Nephrology, Transplantation Center, Department of Nephrology

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045